CLINICAL TRIAL: NCT05960825
Title: Assessment of Two Different Modalities of Maxillary Canine Retraction Assisted With Micro-osteoperforations Versus Injectable Platelet Rich Fibrin: A Comparative Clinical Study
Brief Title: Maxillary Canine Retraction Assisted With Micro-osteoperforations Versus Injectable Platelet Rich Fibrin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 857/140
Record Dates: First submitted 2023-07-15; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Effects of; Movement of Teeth Assiste Wit MOPS and I-prf

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group MOPs (Experimental): Group MOPs : will include 9 patients who willreceive MOPs with maxillary canine retraction that will be performed on intervention sides according to a standardized protocol.
  Interventions: Combination Product: injectable platelet rich fibrin versus microosteoperforation
- Group IMOPS (No Intervention): other side in group which is control group
- Group i-PRF (Experimental): group i-PRF: will include 9 patients receive i-PRF that will be performed on intervention sides according to a standardized protocol
  Interventions: Combination Product: injectable platelet rich fibrin versus microosteoperforation
- group i-PRF2 (No Intervention): other side in group which is control group

INTERVENTIONS:
Combination Product: injectable platelet rich fibrin versus microosteoperforation — injectable platelet rich fibrin which is second product of blood versus microosteoperforation which is surgical procedure
  Arms: Group MOPs; Group i-PRF

SUMMARY:
The present clinical comparative study will be undertaken for assessment of two different modalities of maxillary canine retraction assisted with microosteoperforations versus injectable platelet rich fibrin.

DETAILED DESCRIPTION:
Group I: will include 9 patients who willreceive MOPs with maxillary canine retraction that will be performed on intervention sides according to a standardized protocol.

▪ Group II: will include 9 patients receive i-PRF that will be performed on intervention sides according to a standardized protocol.

ELIGIBILITY:
Inclusion Criteria:

1. An age ranges from 15-22 years.
2. Severe crowding or protrusion requiring 1st premolars extractions followed by symmetrical canine retraction.
3. All permanent teeth present, 3rd molars are excluded.
4. Good oral and general health.
5. No systemic disease/medication that could interfere with OTM.
6. No previous orthodontic treatment.

Exclusion Criteria:

1. Patient diagnosed to have an indication for non-extraction approach.
2. Poor oral hygiene or periodontally compromised patient.
3. Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions.
4. Previous orthodontic treatment.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Direct clinical assessment of the amount of maxillary canine retraction i.e. amount of extraction space closure before and after four months observation period and on every 28 days observation period according to standardized method | 4months
  Direct clinical assessment of the amount of maxillary canine retraction i.e. amount of extraction space closure before and after four months observation and every 28 days period and on every 28 days observation period according to standardized method. 2. Study cast assessment:
  • The amount of maxillary canine retraction on both sides will be measured immediately before starting canine retraction and at each observation interval by using a software for the scanned models according to standardized method

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Result] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053